CLINICAL TRIAL: NCT00335296
Title: The Paradigm IIca/III Trial: PFx Closure System in Subjects With Cryptogenic Stroke, Transient Ischemic Attack, Migraine or Decompression Illness
Brief Title: PFx Closure System in Subjects With Cryptogenic Stroke,Transient Ischemic Attack,Migraine or Decompression Illness(PFO)
Status: Suspended | Phase: Not Applicable | Type: Interventional
Sponsor: Cierra (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA0005/09
Record Dates: First submitted 2006-06-08; First posted 2006-06-09 (Estimated); Last update posted 2007-12-24 (Estimated); Status verified 2007-12

CONDITIONS: Patent Foramen Ovale
Keywords: PFO; Migraine; Stroke; TIA (transient ischemic attack); Decompression Illness
MeSH Terms: conditions — Foramen Ovale, Patent; Migraine Disorders; Stroke; Ischemic Attack, Transient

INTERVENTIONS:
Device: PFx catheter

SUMMARY:
The primary objective of this study is to demonstrate the safety and performance of the PFx Closure System when utilized for patients with PFOs suffering from cryptogenic stroke, transient ischemic attack, migraine or decompression illness.

DETAILED DESCRIPTION:
Patent Foramen Ovale has been implicated in the etiology of paradoxical embolism, cryptogenic stroke, transient ischemic attack, and right to left gas embolism in severe decompression illness. An association between patent foramen ovale and severe migraine headaches has also been reported. Several implantable devices are being used for percutaneous closure of patent foramen ovale; this study uses a non-implantable system to safely effect closure with the application of radiofrequency energy.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years old
* Documented PFO
* Subjects with one or more of the following:cryptogenic stroke, transient ischemic attack, embolism, migraine headaches, decompression illness

Exclusion Criteria:

• Inappropriate anatomy (vascular or cardiac) or inappropriate medical condition for PFO closure and study medications.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-05; Study Completion 2007-12 (Estimated)

PRIMARY OUTCOMES:
PFO closure 6 months post procedure | 6 months

SECONDARY OUTCOMES:
PFO closure at 30 days and 12 months post procedure | 30 days, 12 months
AE event rates for all subjects | 30 days, 6 and 12 months
Migraine severity | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Alec Vahanian, MD, Principal Investigator — Bichat Hospital
Locations (4):
- AZ Middleheim Hospital, Antwerp, Belgium
- France (2):
  - Institut Hospitalier Jacques Carter, Massy
  - Bichat Hospital, Paris
- Cardiovascular Center Frankfurt Sankt katharinen, Frankfurt, Germany